CLINICAL TRIAL: NCT01456845
Title: Estimation of Plasma Free and Total Drug Levels of Rifampicin, Isoniazid and Pyrazinamide in Patients on Antituberculosis Therapy and Its Correlation With Development of Drug Induced Hepatotoxicity
Brief Title: Anti-tuberculosis (TB) Drug Levels and Correlation With Drug Induced Hepatotoxicity
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Head, All India Institute of Medical Sciences
Other Study IDs: SKS/DIH/2011
Record Dates: First submitted 2011-10-20; First posted 2011-10-21 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Hepatitis; Tuberculosis
Keywords: Plasma levels; isoniazid; rifampicin; pyrazinamide; hepatoxicity
MeSH Terms: conditions — Hepatitis; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: Cases - those patients who develop DIH while on regular treatment with anti-TB drugs.
  Controls - patients who do not develop DIH while on regular treatment with anti-TB drugs.

SUMMARY:
The purpose of the study is to estimate plasma drug levels ( free and total drug levels ) of rifampicin and other antituberculosis drugs and compare these drug levels in patients who develop drug induced hepatotoxicity versus those who do not .The study hypothesis is that the ATT drug induced hepatotoxicity is related to free drug levels of rifampicin and other antituberculosis drugs .

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major health problem in both the developing and developed countries because of its resurgence in the immunosuppressed patients. World Health Organization (WHO) in 1993 declared tuberculosis to be a 'global emergency' with more than a third of the world's population infected. Globally 8.9 million new cases of tuberculosis occur annually, of which 1.8 million (20%) occur in India.

Short-course chemotherapy containing isoniazid (INH), rifampicin (RMP) and pyrazinamide (PZA) has proved to be highly effective in the treatment of tuberculosis. One of its adverse effects is hepatotoxicity. It is the most common side effect leading to interruption of therapy. It is associated with mortality of 6-12% if these drugs are continued even after the onset of symptoms. Risk of hepatotoxicity is increased when these drugs are combined.

The time interval between the start of anti-TB drugs and appearance of hepatotoxicity varies from 3 to 135 days. In most cases hepatitis is evident within three months of start of antituberculosis treatment (ATT).

The pathogenesis of drug-induced hepatotoxicity (DIH) is still not entirely clear for most anti TB drugs including rifampicin. Hypersensitivity is a definite possibility. Rifampicin induced hepatitis has been postulated to occur as a part of systemic allergic reaction and due to unconjugated hyperbilirubinaemia as a result of competition with bilirubin for uptake at hepatocyte plasma membrane. DIH caused by rifampicin occurs earlier as compared to isoniazid. While a dose related toxicity may exist, a direct correlation between serum drug levels and hepatotoxicity has not been well reported. Thus the clinical relevance of therapeutic monitoring of serum rifampicin concentrations in managing DIH is still being explored. Rifampicin is highly protein bound and hypoalbuminemia is a known risk factor for DIH ,so free drug levels in plasma has more significance than total drug levels in plasma.

Present study is done to estimate free and total drug levels of rifampicin and other antituberculosis drugs in patients on ATT and to compare it between patients who develop DIH vs those who do not and to assess the predicting ability of these drug levels in the subsequent development of drug induced hepatoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age: patients in the range between 18 to 65 years
* Patients of either gender
* Probable or confirmed cases of TB
* Patients receiving daily antituberculosis drugs

Exclusion Criteria:

* Patients with serological evidence of acute viral hepatitis A, B, C, or E and carriers of HBV and/or HCV
* HIV positive patients
* Presence of chronic liver disease or cirrhosis
* Cognitive dysfunction
* Terminally sick patients and unlikely to survive for 6-9 months
* Concomitant administration of other potentially hepatotoxic drugs(Methotrexate, Phenytoin, phenobarbitone, carbamazepine ,valproate Atenolol, labetalol, Salicylates , allopurinol, quinine, quinidine, fluconazole, cimetidine, ethionamide, verapamil, probenecid, TCA, halothane)
* Chronic alcoholics consuming >48 g/day for more 1 year
* Patients not willing to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects: Patients with diagnosis of pulmonary/extrapulmonary Tuberculosis attending the out-patient department of the All India Institute of Medical Sciences, New Delhi, will form the study population.
  Cases - those patients who develop DIH while on regular treatment with anti-TB drugs Controls - patients who do not develop DIH while on regular treatment with anti-TB drugs
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of plasma levels of isoniazid, rifampicin, pyrazinamide among cases and controls | 21 months

SECONDARY OUTCOMES:
Evaluation of plasma drug levels and its correlation among cases and controls and to assess the ability of these drug levels to predict subsequent development of drug induced hepatoxicity | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD,Ph.D, Principal Investigator — All India Institute of Medical Sciences, New Delhi-110029, India
Locations (1):
- All India Institute of Medical Sciences, New Delhi, India

REFERENCES:
- [Derived] Satyaraddi A, Velpandian T, Sharma SK, Vishnubhatla S, Sharma A, Sirohiwal A, Makharia GK, Sinha S, Biswas A, Singh S. Correlation of plasma anti-tuberculosis drug levels with subsequent development of hepatotoxicity. Int J Tuberc Lung Dis. 2014 Feb;18(2):188-95, i-iii. doi: 10.5588/ijtld.13.0128. PMID 24429311